CLINICAL TRIAL: NCT05366543
Title: Errors of Refraction: Prevalence and Compliance of Wearing Correction Among Primary School Children
Brief Title: Errors of Refraction Among Primary School Children
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Other Study IDs: Paediatric unit
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Error, Refractive
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Visual acuity measurement — Visual acuity will be measured using autorefractometer after cycloplegic eye drops 3 times and glasses will be prescribed for those who are needed.

SUMMARY:
This study will include primary school children to evalute their refraction and follow those who will wear glasses to detect their compliance.

Visual acuity will be measured using autorefractometer after cycloplegic eye drops 3 times and glasses will be prescribed for those who are needed. Follow up of the students to detect their compliance of wearing correction.

ELIGIBILITY:
Inclusion Criteria:

* Primary school student less than 12 years.
* No sensory defect in those children.

Exclusion Criteria:

* Corneal opacity.
* Abnormal fundus lesion.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary school student less than 12 years with no sensory defects in their eyes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity improvement | 3 months
  Measurement of visual acuity after wearing of glasses

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided